CLINICAL TRIAL: NCT05782868
Title: Promoting Well-Being Through Identity Affirmation and Social Connection in TNB Adults: An Expressive Writing Intervention
Brief Title: Expressive Writing Intervention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022-1711; NUR/ACAD SVCS/ACAD SVCS (Other: UW Madison); Protocol Version 11/28/2022 (Other: UW Madison)
Record Dates: First submitted 2023-03-02; First posted 2023-03-24 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Distress, Emotional
Keywords: transgender; nonbinary

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TNB Identity Affirmation (IA) Condition (Experimental): Participants in the IA only intervention condition will receive the same prompt for all four days of writing, a design used in expressive writing interventions to allow for deeper and continued reflection into specific thoughts and emotions.
  Interventions: Other: Expressive writing in response to vignette
- IA + Strengthening Social Connections (SSC) Condition (Experimental): For participants in the IA+SSC condition, participants will complete the IA intervention on the first three days. On the fourth day, participants will be directed to compose a brief letter.
  Interventions: Other: Expressive writing in response to vignette; Other: Letter of Gratitude
- Control Condition (Experimental): Expressive writing assignment, without prompts.
  Interventions: Other: Expressive writing about events of the day

INTERVENTIONS:
Other: Expressive writing in response to vignette — Participants will read a vignette, which describes the experience and response of a young adult who experiences rejection from a close friend after a first disclosure of their gender identity. Participants will then be asked to write in response to three prompts: 1) identify expressions of internalized transphobia in the vignette character, 2) reflect on times the participant has experienced similar feelings, 3) identify thoughts and feelings that promote and support a positive and affirming identity in contrast to negative emotions and thoughts.
  Arms: IA + Strengthening Social Connections (SSC) Condition; TNB Identity Affirmation (IA) Condition
Other: Expressive writing about events of the day — Participants in the control condition will be asked to write about the events of their day and thoughts and feelings that occurred in response to those events.
  Arms: Control Condition
Other: Letter of Gratitude — Participants will be directed to compose a brief letter of gratitude to an individual to whom they have not previously expressed gratitude, and who has provided meaningful and affirming support to them as a TNB person.
  Arms: IA + Strengthening Social Connections (SSC) Condition

SUMMARY:
This study aims to test to what extent an expressive writing intervention may reduce internalized anti-TNB (trans and nonbinary) stigma and promote well-being over time. Trans and/or nonbinary people may take part in this study, and can expect to participate for 3 months.

DETAILED DESCRIPTION:
This study aims to decrease internalized transnegativity and to promote positive and affirming thoughts and emotions related to being transgender/nonbinary through a novel four-day expressive writing intervention. Participants will be trans/nonbinary English-speaking adults (18+) who reside in the US. They will be randomized to one of three study conditions (control, affirming identity, affirming identity + strengthening social connection) and will be enrolled in the study for period of 3 months (baseline, four day intervention, Days 7, 30, and 90 follow up).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* transgender or nonbinary
* access to a phone, computer, and/or device from which they can access the surveys and daily writing session tasks
* ability to read and write English

Exclusion Criteria:

* cisgender individuals
* self-reported severe levels of psychological distress

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2023-09-08 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Assess the feasibility of expressive writing intervention through qualitative data | One week post-baseline
  Collect open-ended text responses to the following question: Considering the logistical and practical side of this study, what was your experience like completing the writing tasks this last week? For example, did you find it easy or challenging to write for the full 20 minutes each session? How was it writing using the device that you did, such as writing in Word and uploading to Qualtrics or writing directly in Qualtrics?
Assess the feasibility of expressive writing intervention by recording the number of attended writing sessions for each participant. | One week post-baseline
  Analyze any differences in number of attended writing sessions for participants by condition, with each participants' attendance score ranging from 0 (none) to 4 (all).
Assess the acceptability of expressive writing intervention through qualitative data | One week post-baseline
  Collect open-ended text responses to the following question:
  Emotionally, what was your experience like completing the writing sessions this last week? Did you notice any changes in your emotional experience over the course of the week?
Effect of missed sessions on Positive and Negative Affect Scale (PANAS) | One week post-baseline
  Participants' total scale scores to the Positive and Negative Affect Scale (PANAS), which can range from 10 to 50, with higher scores indicating greater positive affect (positive affect subscale) and lower scores indicating lower levels of negative affect (negative affect subscale), will be analyzed for their correlations with missed sessions and/or participant attrition, as documented through participant attendance scores, described above.
Assess the fidelity of expressive writing intervention | One week post-baseline
  Analyze participants' writing to assess the degree to which intervention condition writing instructions were followed. Two members of the research team will assess participants' writing and code for the presence of emotion/affect-related words (yes=1, no=0), focus on gender identity (yes=1, no=0), and advice or encouragement offered (yes=1, no=0). Interrater agreement will be assessed.
Amount of time spent writing | One week post-baseline
  To assess fidelity of intervention, participants will be asked to self-report how much time they spent writing each day. Qualtrics data will also be examined to assess how many minutes participants spent in the survey.

SECONDARY OUTCOMES:
Change in resilience as determined by scores on the Brief Resilience Scale (BRS) | Baseline to 3 months
  Using the Brief Resilience Scale, participants will indicate the extent to which they agree with several statements on a scale of 1 to 5, where 1 = strongly disagree and 5 = strongly agree. A higher score indicates lower resilience.
Change in state of depression, anxiety, and stress as determined by their scores on the Depression, Anxiety, and Stress Scale | Baseline to 3 months
  Using the Depression Anxiety Stress Scale (DASS), participants will indicate their negative emotional states of depression, anxiety and stress on a 0-3 scale, with higher scores indicating greater degree of depression, anxiety, or stress.
Change in psychological well-being | Baseline to 3 months
  Using the Psychological Well-Being Scale (PWB), participants will indicate their level of well-being on an 18 item scale, with a range of 1 to 7, where higher scores indicate greater levels of psychological well-being.
Effects of expressive writing intervention on mental health | Baseline to 3 months
  Neuro-QoL short form: Two subscales with 7 (general concerns) and 8 items (fatigue), respectively. Rated on a 1-5 scale, with higher scores indicating lower levels of quality of life in each domain.
Change in Gender Minority Stress and Resilience (GMSR) | Baseline to 3 months
  GMSR: Three subscales with 8 (Pride), 8 (Internalized transphobia), and 5 (community connectedness) items respectively. Rated on a 1-5 scale with higher scores indicating higher levels of pride, internalized transphobia, and community connectedness.
Change in satisfaction with life | Baseline to 3 months
  Participants will indicate agreement with 5 items on a 1 to 7 scale, with higher scores indicating greater satisfaction with life.
Change in perception of social support | Baseline to 3 months
  Using TNB Social Support, participants will report number of contacts, as well as degree of closeness with each contact on a scale of 1 to 7, with higher scores indicating greater perception of social support.

CONTACTS AND LOCATIONS:
Overall Officials: Elliot A Tebbe, PhD, LP, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Researchers may submit a written request to the PI to access de-identified data. The written request should include 1) a short background to describe rationale, 2) a description of the planned analysis, and 3) planned dissemination of findings. The PI reserves the right to approve or disapprove any request. Only de-identified survey data will be shared.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Data will be made available for a period of 5 years post data collection.
Access Criteria: PhD prepared researcher, holds a current appointment in an institution of higher education.